CLINICAL TRIAL: NCT06479096
Title: Four-Week Oral Malodor and Clinical Safety for a Concentrated Cosmetic Mouthwash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS2024OC100108
Record Dates: First submitted 2024-06-24; First posted 2024-06-27 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-08

CONDITIONS: Oral Malodor
MeSH Terms: interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Examiner-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Brush / Espresso Mild Prototype (Experimental): All subjects will receive a marketed fluoride-containing dentifrice and a soft flat trimmed bristled toothbrush to use for the one week wash out period and throughout the study. Subjects will be required to record their daily product use times on a subject diary. After the one week wash out period, subjects subjects will use their assigned mouthwash for the first time at the site under supervision. Subjects will brush their teeth at the site after all assessments are complete. That evening, subjects will brush their teeth and rinse a second time unsupervised. All other twice daily brushing/rinsing will occur unsupervised at home. Subjects will be required to record their daily product use times (brushing and rinsing) on their subject diary.
  Interventions: Other: Brush / Espresso Mild Prototype
- Brush / Espresso Intense Prototype (Experimental): All subjects will receive a marketed fluoride-containing dentifrice and a soft flat trimmed bristled toothbrush to use for the one week wash out period and throughout the study. Subjects will be required to record their daily product use times on a subject diary. After the one week wash out period, subjects subjects will use their assigned mouthwash for the first time at the site under supervision. Subjects will brush their teeth at the site after all assessments are complete. That evening, subjects will brush their teeth and rinse a second time unsupervised. All other twice daily brushing/rinsing will occur unsupervised at home. Subjects will be required to record their daily product use times (brushing and rinsing) on their subject diary.
  Interventions: Other: Brush / Espresso Intense Prototype
- Brush / Fresh Breath Oral Rinse (Active Comparator): All subjects will receive a marketed fluoride-containing dentifrice and a soft flat trimmed bristled toothbrush to use for the one week wash out period and throughout the study. Subjects will be required to record their daily product use times on a subject diary. After the one week wash out period, subjects subjects will use their assigned mouthwash for the first time at the site under supervision. Subjects will brush their teeth at the site after all assessments are complete. That evening, subjects will brush their teeth and rinse a second time unsupervised. All other twice daily brushing/rinsing will occur unsupervised at home. Subjects will be required to record their daily product use times (brushing and rinsing) on their subject diary.
  Interventions: Other: Brush / Fresh Breath Oral Rinse
- Brush / Hydroalcohol (Placebo Comparator): All subjects will receive a marketed fluoride-containing dentifrice and a soft flat trimmed bristled toothbrush to use for the one week wash out period and throughout the study. Subjects will be required to record their daily product use times on a subject diary. After the one week wash out period, subjects subjects will use their assigned mouthwash for the first time at the site under supervision. Subjects will brush their teeth at the site after all assessments are complete. That evening, subjects will brush their teeth and rinse a second time unsupervised. All other twice daily brushing/rinsing will occur unsupervised at home. Subjects will be required to record their daily product use times (brushing and rinsing) on their subject diary.
  Interventions: Other: Brush / Hydroalcohol

INTERVENTIONS:
Other: Brush / Espresso Mild Prototype — Subjects will brush and rinse with their assigned mouthwash twice daily.
  Arms: Brush / Espresso Mild Prototype
Other: Brush / Espresso Intense Prototype — Subjects will brush and rinse with their assigned mouthwash twice daily.
  Arms: Brush / Espresso Intense Prototype
Other: Brush / Fresh Breath Oral Rinse — Subjects will brush and rinse with their assigned mouthwash twice daily.
  Arms: Brush / Fresh Breath Oral Rinse
Other: Brush / Hydroalcohol — Subjects will brush and rinse with their assigned mouthwash twice daily.
  Arms: Brush / Hydroalcohol

SUMMARY:
The objective of this study is to evaluate the safety of the concentrated mouthwash prototypes, and to evaluate the efficacy of the concentrated mouthwash prototypes in the control of oral malodor compared to a comparator mouthwash and a negative control.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and follow the requirements and restrictions of the clinical trial (including willingness to use the assigned study products per instructions, availability on scheduled visit dates and likeliness of completing the clinical trial) based upon research site personnel's assessment;
2. Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial;
3. Able to read and understand the local language (subject is capable of reading the documents);
4. Adequate oral hygiene (i.e., brush teeth daily and exhibit no signs of oral neglect);
5. Adults, 18 years of age and older, in good general and oral health without any known allergy to commercial dental products or cosmetics;
6. Negative pregnancy urine tests (females of child-bearing potential only);

   * For females: Postmenopausal state (i.e. at least 1 year without menses without an alternative medical condition prior to the first study IP administration) or premenopausal/perimenopausal state with an effective means of contraception.
   * For males: No pregnant or lactating spouse or partner at screening and willingness to utilize an acceptable form of birth control with spouse or any potential partner during the study and for 30 days thereafter.
7. Females of childbearing potential must be using a medically acceptable method of birth control for at least one month prior to Visit 1 and agree to continue using this method during their participation in the clinical trial. Medically acceptable forms of birth control that may be used by the subject and/or his/her partner include:

   * Double barrier method (condoms, diaphragm or cervical cap with spermicide),
   * Hormonal prescription contraceptives (i.e., oral, injectable, implanted, patch or vaginal ring hormone therapy)
   * Intrauterine device (IUD)
   * Surgical sterilization (e.g., vasectomy that has been confirmed effective by sperm count check, tubal ligation, hysterectomy and/or bilateral oophorectomy)
   * Abstinence
8. A minimum of 16 uncrowned teeth;
9. At Screening (Visit 1) and before brushing with the assigned study product at Baseline (Visit 2), subjects must provide 2 samples of mouth air, which must have a mean hydrogen sulfide concentration greater than 200ppb. At screening and baseline (pre-brushing), the two samples of mouth air must have a ≤ 500ppb difference in hydrogen sulfide values;
10. At Baseline (Visit 2), before brushing with assigned dentifrice, subjects must provide a breath sample with a mean organoleptic score ≥3.5 across judges;
11. Absence of significant oral soft tissue pathology, periodontitis and active dental caries, based on a visual examination and at the discretion of the Investigator; and
12. Absence of partial dentures, dentures, orthodontic bands, fixed retainers, removable orthodontic appliances.

Exclusion Criteria:

1. Diagnosed with Xerostomia;
2. Suspected alcohol or substance abuse at the discretion of the Investigator (e.g., amphetamines, benzodiazepines, cocaine, marijuana, opiates);
3. Known sensitivity, allergy or contraindications to any investigational product ingredient, oral care products and auxiliary supplies provided for the study;
4. Self-reported smokeless tobacco user including snuff, chewing tobacco, vaping and e-cigarette usage;
5. Females who are pregnant, planning to become pregnant or breastfeeding during the study;
6. Subjects who were previously screened and determined to be ineligible for the study (unless subject previously screen failed for the OralChroma GC and/or organoleptic criteria;
7. Participation in any clinical study investigation within 30 days of Screening visit (Visit 1);
8. Planned surgery during the trial period, 6 months prior to clinic visit 1 or 30 days after the end of study period;
9. Has a compromised immune system;
10. Has any acute or chronic, medical or psychiatric conditions) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgement of the medically qualified investigator, would make the subject inappropriate for entry in this study;
11. Significant, unstable or uncontrolled medical condition which may interfere with subject's participation in the study, at the discretion of the Investigator; and
12. Subjects who are related to those persons involved directly or indirectly with the conduct of this study (i.e., principal Investigator, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson (J&J) subsidiaries, contractors of J&J, and the families of each).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Mean malodor intensity assessed at 60 minutes after product use | After 60 minutes of product use
  Mean malodor intensity will be independently assessed by three odor trained judges 60 minutes after product use on Day 0 using the following scale: 0 = No appreciable odor, 1 = Barely noticeable odor, 2 = Slight but clearly noticeable odor, 3 = Moderate odor, 4 = Strong odor, 5 = Extremely foul odor
Mean malodor intensity assessed at 120 minutes after product use | After 120 minutes of product use
  Mean malodor intensity will be independently assessed by three odor trained judges 120 minutes after product use on Day 0 using the following scale: 0 = No appreciable odor, 1 = Barely noticeable odor, 2 = Slight but clearly noticeable odor, 3 = Moderate odor, 4 = Strong odor, 5 = Extremely foul odor
Mean malodor intensity assessed at 180 minutes after product use | After 180 minutes of product use
  Mean malodor intensity will be independently assessed by three odor trained judges 180 minutes after product use on Day 0 using the following scale: 0 = No appreciable odor, 1 = Barely noticeable odor, 2 = Slight but clearly noticeable odor, 3 = Moderate odor, 4 = Strong odor, 5 = Extremely foul odor
Mean malodor intensity assessed at 240 minutes after product use | After 240 minutes of product use
  Mean malodor intensity will be independently assessed by three odor trained judges 240 minutes after product use on Day 0 using the following scale: 0 = No appreciable odor, 1 = Barely noticeable odor, 2 = Slight but clearly noticeable odor, 3 = Moderate odor, 4 = Strong odor, 5 = Extremely foul odor
Mean malodor intensity assessed at 12 hours after product use on Day 7 | After 12 hours of product use on Day 7
  Mean malodor intensity will be independently assessed by three odor trained judges 12 hours after product use on Day 7 using the following scale: 0 = No appreciable odor, 1 = Barely noticeable odor, 2 = Slight but clearly noticeable odor, 3 = Moderate odor, 4 = Strong odor, 5 = Extremely foul odor
Mean malodor intensity assessed at 12 hours after product use on Day 21 | After 12 hours of product use on Day 21
  Mean malodor intensity will be independently assessed by three odor trained judges 12 hours after product use on Day 21 using the following scale: 0 = No appreciable odor, 1 = Barely noticeable odor, 2 = Slight but clearly noticeable odor, 3 = Moderate odor, 4 = Strong odor, 5 = Extremely foul odor

SECONDARY OUTCOMES:
Total volatile sulfur compounds (VSC) concentration assessed at 60 minutes after product use on Day 0 | After 60 minutes of product use
  Two mouth air sample will be evaluated 60 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the total VSC concentration in breath (hydrogen sulfide, methyl mercaptan, and methyl sulfide) in the range of 50- 2400ppb.
Total volatile sulfur compounds (VSC) concentration assessed at 120 minutes after product use on Day 0 | After 120 minutes of product use
  Two mouth air sample will be evaluated 120 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the total VSC concentration in breath (hydrogen sulfide, methyl mercaptan, and methyl sulfide) in the range of 50- 2400ppb.
Total volatile sulfur compounds (VSC) concentration assessed at 180 minutes after product use on Day 0 | After 180 minutes of product use
  Two mouth air sample will be evaluated 180 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the total VSC concentration in breath (hydrogen sulfide, methyl mercaptan, and methyl sulfide) in the range of 50- 2400ppb.
Total volatile sulfur compounds (VSC) concentration assessed at 240 minutes after product use on Day 0 | After 240 minutes of product use
  Two mouth air sample will be evaluated 240 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the total VSC concentration in breath (hydrogen sulfide, methyl mercaptan, and methyl sulfide) in the range of 50- 2400ppb.
Total volatile sulfur compounds (VSC) concentration assessed at 12 hours after product use on Day 7 | After 12 hours of product use on Day 7
  Two mouth air sample will be evaluated 12 hours after product use on Day 7 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the total VSC concentration in breath (hydrogen sulfide, methyl mercaptan, and methyl sulfide) in the range of 50- 2400ppb.
Total volatile sulfur compounds (VSC) concentration assessed at 12 hours after product use on Day 21 | After 12 hours of product use on Day 21
  Two mouth air sample will be evaluated 12 hours after product use on Day 21 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the total VSC concentration in breath (hydrogen sulfide, methyl mercaptan, and methyl sulfide) in the range of 50- 2400ppb.
Hydrogen sulfide concentration assessed at 60 minutes after product use on Day 0 | After 60 minutes of product use on Day 0
  Two mouth air sample will be evaluated 60 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the hydrogen sulfide concentration in the breath in the range of 50- 2400ppb.
Hydrogen sulfide concentration assessed at 120 minutes after product use on Day 0 | After 120 minutes of product use on Day 0
  Two mouth air sample will be evaluated 120 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the hydrogen sulfide concentration in the breath in the range of 50- 2400ppb.
Hydrogen sulfide concentration assessed at 180 minutes after product use on Day 0 | After 180 minutes of product use on Day 0
  Two mouth air sample will be evaluated 180 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the hydrogen sulfide concentration in the breath in the range of 50- 2400ppb.
Hydrogen sulfide concentration assessed at 240 minutes after product use on Day 0 | After 240 minutes of product use on Day 0
  Two mouth air sample will be evaluated 240 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the hydrogen sulfide concentration in the breath in the range of 50- 2400ppb.
Hydrogen sulfide concentration assessed at 12 hours after product use on Day 7 | After 12 hours of product use on Day 7
  Two mouth air sample will be evaluated 12 hours after product use on Day 7 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the hydrogen sulfide concentration in the breath in the range of 50- 2400ppb.
Hydrogen sulfide concentration assessed at 12 hours after product use on Day 21 | After 12 hours of product use on Day 21
  Two mouth air sample will be evaluated 12 hours after product use on Day 21 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the hydrogen sulfide concentration in the breath in the range of 50- 2400ppb.
Methyl mercaptan concentration assessed at 60 minutes after product use on Day 0 | After 60 minutes of product use on Day 0
  Two mouth air sample will be evaluated 60 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the methyl mercaptan concentration in the breath in the range of 50- 2400ppb.
Methyl mercaptan concentration assessed at 120 minutes after product use on Day 0 | After 120 minutes of product use on Day 0
  Two mouth air sample will be evaluated 120 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the methyl mercaptan concentration in the breath in the range of 50- 2400ppb.
Methyl mercaptan concentration assessed at 180 minutes after product use on Day 0 | After 180 minutes of product use on Day 0
  Two mouth air sample will be evaluated 180 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the methyl mercaptan concentration in the breath in the range of 50- 2400ppb.
Methyl mercaptan concentration assessed at 240 minutes after product use on Day 0 | After 240 minutes of product use on Day 0
  Two mouth air sample will be evaluated 240 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the methyl mercaptan concentration in the breath in the range of 50- 2400ppb.
Methyl mercaptan concentration assessed at 12 hours after product use on Day 7 | After 12 hours of product use on Day 7
  Two mouth air sample will be evaluated 12 hours after product use on Day 7 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the methyl mercaptan concentration in the breath in the range of 50- 2400ppb.
Methyl mercaptan concentration assessed at 12 hours after product use on Day 21 | After 12 hours of product use on Day 21
  Two mouth air sample will be evaluated 12 hours after product use on Day 21 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the methyl mercaptan concentration in the breath in the range of 50- 2400ppb.
Methyl sulfide concentration assessed at 60 minutes after product use on Day 0 | After 60 minutes of product use on Day 0
  Two mouth air sample will be evaluated 60 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the methyl mercaptan concentration in the breath in the range of 50- 2400ppb.
Methyl sulfide concentration assessed at 120 minutes after product use on Day 0 | After 120 minutes of product use on Day 0
  Two mouth air sample will be evaluated 120 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the methyl mercaptan concentration in the breath in the range of 50- 2400ppb.
Methyl sulfide concentration assessed at 180 minutes after product use on Day 0 | After 180 minutes of product use on Day 0
  Two mouth air sample will be evaluated 180 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the methyl mercaptan concentration in the breath in the range of 50- 2400ppb.
Methyl sulfide concentration assessed at 240 minutes after product use on Day 0 | After 240 minutes of product use on Day 0
  Two mouth air sample will be evaluated 240 minutes after product use on Day 0 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the methyl mercaptan concentration in the breath in the range of 50- 2400ppb.
Methyl sulfide concentration assessed at 12 hours after product use on Day 7 | After 12 hours of product use on Day 7
  Two mouth air sample will be evaluated 12 hours after product use on Day 7 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the methyl mercaptan concentration in the breath in the range of 50- 2400ppb.
Methyl sulfide concentration assessed at 12 hours after product use on Day 21 | After 12 hours of product use on Day 21
  Two mouth air sample will be evaluated 12 hours after product use on Day 21 using the Oral Chroma Halitosis Measuring instrument, a portable gas chromatograph with a highly sensitive semiconductor gas detector that will determine the methyl mercaptan concentration in the breath in the range of 50- 2400ppb.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Milleman, DDS, Principal Investigator — Salus Research Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu